CLINICAL TRIAL: NCT05469048
Title: Near Patient Molecular Testing in Sepsis
Acronym: NEPTUNE
Status: Completed | Type: Observational
Sponsor: Immunexpress (Industry)
Collaborators: Rush University Medical Center (Other); Grady Memorial Hospital (Other); University of Southern California (Other)
Responsible Party: Sponsor
Other Study IDs: NEPTUNE IXP-181
Record Dates: First submitted 2022-07-15; First posted 2022-07-21 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Sepsis; Systemic Inflammatory Response Syndrome
MeSH Terms: conditions — Sepsis; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples collected in PAXgene RNA tubes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients sepsis suspected: Patients suspected of sepsis and admitted to ICU

SUMMARY:
The purpose of the study is to evaluate the real-time performance of a new host response test (SeptiCyte RAPID) for differentiating sepsis from non-infection/systemic inflammatory response syndrome among patients suspected of sepsis within the first 24 hours of intensive care unit (ICU) admission.

DETAILED DESCRIPTION:
The ability of SeptiCyte RAPID to differentiate sepsis from infection-negative systemic inflammation will be determined using retrospective physician diagnosis performed by an external panel of three physicians not involved with the care of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old on the date of ICU admission
2. Systemic Inflammatory Response Syndrome (SIRS) present, as defined by the presence of two or more of the following:

   1. Temperature > 38°C or < 36°C
   2. Heart Rate > 90 beat/min
   3. Tachypnea > 20/min or PaCO2 < 32 mmHg
   4. WBC count > 12 000/mm3 or < 4 000/mm3 or > 10% immature neutrophils (bands)
3. Consent to study inclusion, either by patient or legal surrogate before study-related sample processing
4. Study sample collection within 24 hours of ICU admission order

Exclusion Criteria:

1. Age less than 18 years old on the day of ICU admission
2. No order to admit to ICU
3. Not physically admitted to ICU
4. Commencement of non-prophylactic antibiotics ≥ 24 hours prior to ICU admission
5. Study sample collection > 24 hours from ICU admission order
6. No clinical cultures or serologic tests obtained when sepsis was suspected
7. Elective cardiac surgery patients with an expected duration in ICU of less than 24 hours
8. Transfer from another ICU where subject was admitted for ≥ 24 hours.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suspected of sepsis, admitted to an Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Real-time evaluation of the diagnostic accuracy of SeptiCyte RAPID in differentiating sepsis from non-infectious systemic inflammation in patients admitted to the ICU. | Time for enrollment, process samples, and collect data, an average of 1 year
  Percentage of correctly identified patients with sepsis or non-infectious systemic inflammation using SeptiCyte RAPID compared to clinical assessments using routine clinical, laboratory, and other findings.

SECONDARY OUTCOMES:
Comparison of diagnostic accuracy between SeptiCyte RAPID and up to 15 other clinical parameters in differentiating sepsis from non-infectious systemic inflammation in patients admitted to the ICU. | Time for enrollment, process samples, and collect data, an average of 1 year
  Multi-parametric model to compare diagnostic accuracy between SeptiCyte RAPID alone or in combination with up to 15 other clinical parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Davis, MD, PhD, MHA, Study Director — Immunexpress
Locations (3):
- United States (3):
  - Keck Hospital of University of Southern California (USC) and Los Angeles County and USC Medical Center, Los Angeles, California
  - Grady Memorial Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Balk R, Esper AM, Martin GS, Miller RR 3rd, Lopansri BK, Burke JP, Levy M, Opal S, Rothman RE, D'Alessio FR, Sidhaye VK, Aggarwal NR, Greenberg JA, Yoder M, Patel G, Gilbert E, Parada JP, Afshar M, Kempker JA, van der Poll T, Schultz MJ, Scicluna BP, Klein Klouwenberg PMC, Liebler J, Blodget E, Kumar S, Navalkar K, Yager TD, Sampson D, Kirk JT, Cermelli S, Davis RF, Brandon RB. Validation of SeptiCyte RAPID to Discriminate Sepsis from Non-Infectious Systemic Inflammation. J Clin Med. 2024 Feb 20;13(5):1194. doi: 10.3390/jcm13051194. PMID 38592057